CLINICAL TRIAL: NCT00279916
Title: Short Term Relief of Eustachian Tube Dysfunction and Serous Otitis Media Using Intranasal Steroid Sprays: a Randomized Placebo-controlled Study
Brief Title: Short Term Relief of Eustachian Tube Dysfunction and Serous Otitis Media Using Intranasal Steroid Sprays
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Laura Orvidas, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 103-04; IST4008 (Other Grant/Funding Number: Sanofi-Aventis US, LLC)
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Otitis Media, Serous; Negative Middle Ear Pressure; Rhinitis; Otitis Media With Effusion; Otitis Media, Secretory
MeSH Terms: conditions — Otitis Media with Effusion; Rhinitis | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triamcinolone acetonide (Active Comparator): Triamcinolone acetonide nasal spray; Subjects aged 12 years or older received 2 metered sprays in each nostril once daily (55 micrograms/spray) (total daily dose 220 micrograms) for 6 weeks duration.
  Subjects younger than 12 years old received received 1 metered spray in each nostril once daily (55 micrograms/spray) (total daily dose 110 micrograms) for 6 weeks duration.
  Interventions: Drug: Triamcinolone acetonide nasal spray
- Placebo (Sham Comparator): Placebo nasal spray; Subjects aged 12 years or older received an aqueous solution lacking triamcinolone, 2 metered sprays in each nostril once daily for 6 weeks duration.
  Subjects younger than 12 years old received received 1 metered spray of placebo solution in each nostril once daily for 6 weeks duration.
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Triamcinolone acetonide nasal spray — Subjects aged 12 years or older received 2 metered sprays in each nostril once daily (55 micrograms/spray) (total daily dose 220 micrograms).
  Subjects younger than 12 years old received received 1 metered spray in each nostril once daily (55 micrograms/spray) (total daily dose 110 micrograms).
  Other Names: Nasacort AQ
  Arms: Triamcinolone acetonide
Drug: Placebo nasal spray — Subjects aged 12 years or older received an aqueous solution lacking triamcinolone, 2 metered sprays in each nostril once daily.
  Subjects younger than 12 years old received received 1 metered spray of placebo solution in each nostril once daily.
  Arms: Placebo

SUMMARY:
We hypothesize that intranasal steroid application will have a beneficial therapeutic effect in adults with regard to resolution of serous otitis media and/or negative middle ear pressure, as compared to placebo. We further hypothesize that the rate of spontaneous short-term resolution of otitis media wit effusion in adults treated with placebo will be relatively low (minority of patients).

DETAILED DESCRIPTION:
Newer intranasal steroid preparations are generally safe with relatively few side effects as demonstrated in large studies dealing with allergic rhinitis.

Eustachian Tube Dysfunction (ETD) primarily refers to an absent or inadequate ability to open the eustachian tube. The term Serous Otitis Media (SOM) generally referring to an accumulation of fluid within the middle ear space, in absence of signs indicating acute infection. Commonly, this can result in a conductive hearing loss due to restriction of tympanic membrane mobility. Negative Middle Ear Pressure (NMEP) is often a precursor to the development of SOM, and has it's own effect on the acoustic properties of the middle ear, also resulting in conductive hearing loss.

Due to the lack of a single accepted medical intervention to deal with ETD and the general benign nature of this condition, it is common practice for some physicians to take a "wait and see" initial approach when this clinical entity is encountered in lieu of prescribing unproved medications. It is generally accepted that some patients with Negative Middle Ear Pressure (NMEP) and/or Serous Otitis Media (SOM) will undergo spontaneous resolution of symptoms, yet the exact resolution rates are not clearly defined.

The purpose of this double-blind, randomized study of either triamcinolone acetonide nasal spray or a sham placebo nasal spray for 6 weeks is to determine if there is improvement in a test of middle ear pressure. Neither the subjects nor the Investigator will know which of the two treatments is being used until the end of the study.

Resolution of ETD symptoms will be measured by changes in the tympanogram, a test to measure pressure within the middle ear. This measurement will be taken at baseline and after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 0-18 years
* Patients with serous otitis media and/or negative middle ear pressure as documented by otoscopic examination and tympanometry will be considered for enrollment
* Pregnant

Exclusion Criteria:

* Unwilling to discontinue breast feeding, when applicable
* Active upper respiratory infection
* Nasopharyngeal mass
* Chronic infectious otitis media
* Cholesteatoma
* Acute infectious otitis media
* History of otologic surgery other than placement of a pressure equalizer tube in the affected ear
* History of radiation therapy to the head and neck region
* Neuromuscular disease
* Cystic fibrosis
* Immunodeficiency
* Mucociliary disorders
* Craniofacial disorders/syndromes
* Cleft palate
* Development delay and/or symptoms suggestive of perilymph fistula

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura J. Orvidas, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gluth MB, McDonald DR, Weaver AL, Bauch CD, Beatty CW, Orvidas LJ. Management of eustachian tube dysfunction with nasal steroid spray: a prospective, randomized, placebo-controlled trial. Arch Otolaryngol Head Neck Surg. 2011 May;137(5):449-55. doi: 10.1001/archoto.2011.56. PMID 21576556
- [Derived] Mulvaney CA, Galbraith K, Webster KE, Rana M, Connolly R, Tudor-Green B, Marom T, Daniel M, Venekamp RP, Schilder AG, MacKeith S. Topical and oral steroids for otitis media with effusion (OME) in children. Cochrane Database Syst Rev. 2023 Dec 13;12(12):CD015255. doi: 10.1002/14651858.CD015255.pub2. PMID 38088821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from the patients seen at the Mayo Clinic Department of Otorhinolaryngology (Ears, Nose and Throat) in Rochester, Minnesota. Enrollment occurred from 09/01/2005 through 12/31/2008.
Groups:
- Triamcinolone Acetonide: Triamcinolone acetonide nasal spray; Subjects aged 12 years or older received 2 metered sprays in each nostril once daily (55 micrograms/spray) (total daily dose 220 micrograms) for 6 weeks duration.
  Subjects younger than 12 years old received 1 metered spray in each nostril once daily (55 micrograms/spray) (total daily dose 110 micrograms) for 6 weeks duration.
- Placebo: Placebo nasal spray; Subjects aged 12 years or older received an aqueous solution lacking triamcinolone, 2 metered sprays in each nostril once daily for 6 weeks duration.
  Subjects younger than 12 years old received 1 metered spray of placebo solution in each nostril once daily for 6 weeks duration.
Period: Overall Study
Arm/Group | Triamcinolone Acetonide | Placebo
Started | 45 | 46
Completed | 38 | 41
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone Acetonide | Placebo | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 18 | 34
  Between 18 and 65 years | 18 | 12 | 30
  >=65 years | 11 | 16 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (28.4) | 42.0 (30.8) | 41.7 (29.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 16 | 46
  Male | 15 | 30 | 45
Tympanogram type in worst ear [Number; unit: participants]
  A; peak pressure under -100 kPa | 0 | 0 | 0
  B; non-peaked or flat pressure | 17 | 16 | 33
  C; peaked pressure greater than -100 kPa | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Complete Normalization of Abnormal Tympanometry, Regardless of Additional Treatment
Description: Number of subjects with resolution of eustachian tube dysfunction symptoms, as determined by the change in tympanogram type in both ears from an initial Type B or C result to Type A result at 6 weeks. Type A; peaked pressure measurement under -100 kilo Pascals (kPa). Type B; non-peaked, or flat tympanogram, Type C; peaked pressure measurements more negative than -100 kPa. A Pascal is a unit used to quantify internal pressure.
Time Frame: 6 weeks
Population: Number of participants is based on those who completed the study and who had a follow-up tympanogram. 37 of the subjects randomized to Triamcinolone acetonide nasal spray and 37 of the subjects randomized to placebo had a follow-up tympanogram at 6 weeks.
Measure: Number; unit: participants
Arm/Group | Triamcinolone Acetonide | Placebo
Number analyzed (Participants) | 37 | 37
participants | 7 | 12
Statistical Analysis 1: Comparison: Triamcinolone Acetonide vs Placebo; Test type: Superiority; p = 0.18, Chi-squared

2. Secondary Outcome: Complete Normalization of Abnormal Tympanometry Considering the Subjects Who Took Additional Treatment as Having Incomplete Resolution
Description: For this outcome measure, the subjects treated with antibiotics or oral decongestants while enrolled in the study were handled as having treatment failures. For this outcome measure, subjects with complete normalization of abnormal tympanometry at 6 weeks had a Type A tympanogram and did not take antibiotics, oral decongestants, nasal spray or a combination.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Triamcinolone Acetonide | Placebo
Number analyzed (Participants) | 37 | 37
participants | 5 | 9
Statistical Analysis 1: Comparison: Triamcinolone Acetonide; Test type: Superiority; p = 0.24, Chi-squared

3. Secondary Outcome: Per-Ear Treatment Outcome
Description: Initial Tympanogram Type at baseline was compared to Follow-Up Tympanogram Type at 6 weeks. Type A is considered to be normal. Type A; peaked pressure measurement under -100 kilo Pascals (kPa). Type B; non-peaked, or flat tympanogram, Type C; peaked pressure measurements more negative than -100 kPa. A Pascal is a unit used to quantify internal pressure.
Time Frame: baseline, 6 weeks
Population: as for outcome 1
Measure: Number; unit: ears
Arm/Group | Triamcinolone Acetonide | Placebo
Number analyzed (Participants) | 37 | 37
ears
  Initial Tympanogram of Type B or C | 55 | 57
  6 weeks Complete Normalization (Type A) | 12 | 20

4. Secondary Outcome: Number of Subjects With Change in Symptom Frequency and Severity - Fullness or Pressure in Ears
Description: As measured by the Eustachian Tube Dysfunction Questionnaire. The questionnaire had 5 symptoms with a Frequency Rating from 1=Never to 5=Constantly, and Severity rating from 1=None at all to 5=Maximum severity. The change in frequency and severity ratings were categorized as same, better, or worse.
Time Frame: baseline, 6 weeks
Population: Number of participants is based on those who completed the study and who completed a baseline and a follow-up questionnaire. 38 of the subjects randomized to Triamcinolone acetonide nasal spray and 40 of the subjects randomized to placebo had a baseline and follow-up questionnaire at 6 weeks.
Measure: Number; unit: participants
Arm/Group | Triamcinolone Acetonide | Placebo
Number analyzed (Participants) | 38 | 40
participants
  Frequency - Better | 11 | 18
  Frequency - Same | 17 | 17
  Frequency - Worse | 10 | 5
  Severity - Better | 13 | 18
  Severity - Same | 14 | 13
  Severity - Worse | 11 | 9

5. Secondary Outcome: Number of Subjects With Change in Symptom Frequency and Severity - Pain in Ears
Description: as for outcome 4
Time Frame: baseline, 6 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Triamcinolone Acetonide | Placebo
Number analyzed (Participants) | 38 | 40
participants
  Frequency - Better | 11 | 8
  Frequency - Same | 17 | 23
  Frequency - Worse | 10 | 9
  Severity - Better | 9 | 6
  Severity - Same | 19 | 25
  Severity - Worse | 10 | 9

6. Secondary Outcome: Number of Subjects With Change in Symptom Frequency and Severity - Plugged Sensation in Ears
Description: as for outcome 4
Time Frame: baseline, 6 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Triamcinolone Acetonide | Placebo
Number analyzed (Participants) | 38 | 40
participants
  Frequency - Missing | 0 | 1
  Frequency - Better | 10 | 14
  Frequency - Same | 13 | 21
  Frequency - Worse | 15 | 4
  Severity - Missing | 0 | 1
  Severity - Better | 15 | 14
  Severity - Same | 8 | 16
  Severity - Worse | 15 | 9

7. Secondary Outcome: Number of Subjects With Change in Symptom Frequency and Severity - Popping Sensation in Ears
Description: as for outcome 4
Time Frame: baseline, 6 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Triamcinolone Acetonide | Placebo
Number analyzed (Participants) | 38 | 40
participants
  Frequency - Missing | 0 | 1
  Frequency - Better | 11 | 8
  Frequency - Same | 14 | 18
  Frequency - Worse | 13 | 13
  Severity - Missing | 0 | 2
  Severity - Better | 9 | 6
  Severity - Same | 17 | 19
  Severity - Worse | 12 | 13

8. Secondary Outcome: Number of Subjects With Change in Symptom Frequency and Severity - Dampened Hearing/Loss Worse Than Usual
Description: as for outcome 4
Time Frame: baseline, 6 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Triamcinolone Acetonide | Placebo
Number analyzed (Participants) | 38 | 40
participants
  Frequency - Missing | 0 | 1
  Frequency - Better | 16 | 16
  Frequency - Same | 14 | 15
  Frequency - Worse | 8 | 8
  Severity - Missing | 0 | 1
  Severity - Better | 15 | 14
  Severity - Same | 13 | 15
  Severity - Worse | 10 | 10

ADVERSE EVENTS:
Arm/Group | Triamcinolone Acetonide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/41
Other Adverse Events (participants affected / at risk) | 0/45 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No